CLINICAL TRIAL: NCT06876493
Title: Comparison of the Effects of Whole Body Vibration Training and Aerobic Exercise on Premanstrual Syndrome in Young Women on a Routine Dietary Intake: a Randomised Controlled Trial
Brief Title: Comparison of the Effects of Whole Body Vibration Training and Aerobic Exercise on Premanstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Derya Azim, Asst. Prof., Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-242
Record Dates: First submitted 2025-02-28; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-08

CONDITIONS: Exercise; Whole Body Vibration
Keywords: Whole Body Vibration; Exercise; Premanstrual Syndrome
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic Exercise Programme (Experimental): The aerobic exercise programme was shown to female students with premenstrual syndrome on the first day by the researcher (D.A.) at the sports centre. Participants were advised to drink water and wear running shoes during exercise. Warm-up exercises were performed for 10 minutes before the exercise. Exercise intensity was determined by the Karvonen formula (HRmax=220-age, HRR=HRmax-HR rest, 60% THR=(0.60xHRR)+HR rest). According to the pulse rate of the exercise, pulse values are monitored on the treadmill and km/hour speeds are adjusted according to pulse values. The exercise programme started with low aerobic exercise intensity on the treadmill, gradually increased at 5-minute intervals and completed at 40-60% of the heart rate, and finally 5 minutes of light stretching movements were performed to return to the initial state. In the following sessions, the participants performed the exercise programmes individually at the sports centre for 45 minutes (10 min warm-up, 30 min walk
  Interventions: Other: Aerobic Exercise Programme
- Whole Body Vibration Training Programme (Experimental): The WBV programme used a frequency of 25 Hz and an amplitude of 2 mm (low amplitude). The Power Plate® (pro5TM) machine provided the device's vibration. This device provides a three-plane oscillatory motion. The programme lasted eight weeks and was performed three days a week. There was at least one day's rest between each session. Before and after each vibration, stretching exercises (warm-up and cool-down programme) were performed for 5 minutes, particularly for the quadriceps and trunk extensors. The participants exercised in three different positions on the vibration platform: 1. Squat position: The knee angle was set at 120° to reduce the transmission of vibrations to the upper body (spine and head) and to increase the load on the leg muscles. 2. Bridge position: Participants stood statically in the bridge position with the soles of both feet on the platform. 3. Push-up position: Participants stood statically in the push-up position with both hands on the platform.
  Interventions: Other: Whole Body Vibration Training Programme

INTERVENTIONS:
Other: Aerobic Exercise Programme — The aerobic exercise programme was shown to female students with premenstrual syndrome on the first day by the researcher (D.A.) at the sports centre. Participants were advised to drink water and wear running shoes during exercise. Warm-up exercises were performed for 10 minutes before the exercise. Exercise intensity was determined by the Karvonen formula (HRmax=220-age, HRR=HRmax-HR rest, 60% THR=(0.60xHRR)+HR rest). .According to the pulse rate of the exercise, pulse values are monitored on the treadmill and km/hour speeds are adjusted according to pulse values. The exercise programme started with low aerobic exercise intensity on the treadmill, gradually increased at 5-minute intervals and completed at 40-60% of the heart rate, and finally 5 minutes of light stretching movements were performed to return to the initial state. In the following sessions, the participants performed the exercise programmes individually at the sports centre for 45 minutes (10 min warm-up, 30 min walk,
  Arms: Aerobic Exercise Programme
Other: Whole Body Vibration Training Programme — The WBV programme used a frequency of 25 Hz and an amplitude of 2 mm (low amplitude). The Power Plate® (pro5TM) machine provided the device's vibration. This device provides a three-plane oscillatory motion. The programme lasted eight weeks and was performed three days a week. There was at least one day's rest between each session. Before and after each vibration, stretching exercises (warm-up and cool-down programme) were performed for 5 minutes, particularly for the quadriceps and trunk extensors
  Arms: Whole Body Vibration Training Programme

SUMMARY:
Aim: The aim of the study was to compare the effects of whole body vibration training (WBVT) and aerobic exercise on premenstrual syndrome in young women with routine dietary intake.

DETAILED DESCRIPTION:
Methods: A prospective, randomised, pre-post-test, single-blind, controlled study was conducted in 34 women diagnosed with PMS. Participants were randomly assigned into three groups: the Aerobic Exercise Group (AEG, n=11), the Whole-Body Vibration Training Group (WBVT, n=11), and the Control Group (CG, n=12). Participants in the AEG performed 45-minute exercise sessions (10 minutes warm-up, 30 minutes walk, 5 minutes cool down) three times a week for eight weeks. The WBV program was conducted using a 25 Hz frequency and a 2 mm low amplitude on the Power Plate® (pro5TM) machine, which provides three-plane oscillatory motion. The program lasted eight weeks, with sessions held three days a week, ensuring at least one rest day between sessions. The control group was asked to continue their daily life routines. Dietary intake of all participants was monitored, and those with different diets were excluded from the study. Premenstrual Syndrome Questionnaire (PMSS) was used to evaluate PMS symptoms and Visual Analogue Scale (VAS) was used to evaluate pain.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5-25
* Score over 110 points on the PMS questionnaire
* To be between the ages of 18-35
* Sedentary women
* Having a regular menstrual cycle (24-35 days)

Exclusion Criteria:

* Diagnosed with eating disorder
* Taking nutritional supplements before the last three cycles
* DM, thyroid and liver kidney disorders
* Endocrine drug use
* Has undergone orthopedic surgery within the last 6 months
* With a neurological diagnosis
* With limited range of motion
* Diagnosed with cardiovascular and cardiopulmonary system disorders
* Diagnosed with women's health and diseases such as polycystic ovary syndrome, endometriosis
* Oral contraceptive users
* Psychiatric diagnosis
* Smoking
* Diagnosed with Amenorrhea
* Following a regular diet
* During pregnancy and lactation

Ages: 18 Years to 32 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — woman
Enrollment: 34 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS) | baseline-8 week
  The scale, which was developed and a validity and reliability study was carried out by Gençdoğan to measure premenstrual symptoms and determine their severity, consists of 44 items in 5-point Likert type. PMSS total score' is obtained by summing the scores obtained from these sub-dimensions. The lowest score that can be obtained from the scale is 44 and the highest score is 220. A high score indicates that the intensity of PMS symptoms is high. When the results of the PMSS are evaluated, it is decided whether PMS is present or absent according to whether the total and subscale scores exceed 50% of the highest score that can be obtained
Visual Analogue Scale (VAS) | baseline-8 week
  In all groups, the pain intensity of the patients will be graded between 0 (no pain) and 10 (unbearable pain) using VAS. VAS is a very common scale used for pain assessment in daily practice and pain averages ranging from 0 to 10 are given in this assessment. Accordingly, '0' indicates the absence of pain, while a mean VAS value of 1-4 indicates mild pain, 5-6 indicates moderate pain and 7-10 indicates severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Derya Azim, Bandırma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author, upon reasonable request